CLINICAL TRIAL: NCT06815198
Title: Pulsed Eco Doppler for the Study of Polmonal Discharge Velocity: Pilot/Explorative Study
Brief Title: Pulsed Eco Doppler for Polmonal Discharge Velocity
Acronym: VeLung
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: VeLung
Record Dates: First submitted 2024-11-28; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-10

CONDITIONS: LUNG
Keywords: PULSED ECO DOPPLER, LUNG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: The first group will include subjects without pulmonary disease who will be admitted to the pulmonology outpatient clinic, where they will undergo respiratory function and ultrasound tests simultaneously by two operators respectively
- Group 2: The second group includes three subgroups of patients:
  2a) Patients with chronic respiratory diseases referred to the Respiratory Diseases Unit of this Polyclinic classified according to the type of disease: COPD, Idiopathic Pulmonary Fibrosis, Pneumonia, Asthma in good control and exacerbation, neuromuscular diseases, ARDS (group2a).
  2b) The patients without pulmonary diseases and undergoing elective surgery mechanically ventilated (group2b).
  2c) The patients with pulmonary diseases undergoing surgery in the operating room surgery and/or admitted to the Multipurpose Intensive Care Unit and Respiratory Intensive Care Unit of this Polyclinic undergoing mechanical ventilation, categorized according to the type of lung disease specified in the previous point(group2c).

SUMMARY:
Chest ultrasound is increasingly being used in the diagnosis and management of the respiratory patient. With ultrasound, ultrasound artifacts representing the lung during inspiration and during exhalation are visualized and analyzed. During inspiration, the lung inflates with air while when exhaling, the lung empties. These two phases are visualized on ultrasound with a sliding motion of the pleural line, which represents the margin of the lung.

The aim of the study is to identify the speed of filling and emptying of the lung by studying the characteristics of the pulsed Doppler wave to measure the speed of lung sliding as the significance of this finding has not yet been clarified. In both healthy subjects and patients with lung disease, it is not known whether there is a correlation between velocity measured by the Doppler wave with the main data recorded by a mechanical ventilator or spirometer.

DETAILED DESCRIPTION:
In the context of trauma, lung ultrasound has proven to be an indispensable tool for identifying pneumothorax. Two ultrasound signs confirm the presence of pnx : the absence of pleural gliding and the finding of the lung point, which is the point where the partially collapsed lung regains contact with the pleural leaflets. However, it is not always easy to be able to detect these two signs especially in the field of urgency-emergency, which is why the authors of the extended focused assessment sonography for trauma (EFAST) proposed to include in the extended ultrasound study the use of Color Doppler by attributing the terms "power slide" to confirm the presence of pleural motion and be able to exclude pneumothorax. The use of Color Doppler has always been used for the identification of blood vessels based on the movement of blood flow. The unusual use of Color Doppler in this context finds its rationale in the physical principle that the Doppler wave senses the motion of approaching and receding from the probe regardless of whether the insonated object is a vascular structure or a biological tissue.

The literature shows that pulmonary Doppler was used in a pilot study to analyze pulmonary vessels in healthy individuals and compare it with individuals in whom pulmonary embolism was established by CT angiography.

In contrast, the use of pulsed Doppler or tissue Doppler to measure the rate of lung parenchyma sliding has not yet been investigated.

Therefore, it is unclear whether pulsed Doppler can measure the velocity of lung gliding and whether this measurement correlates with flow values collected during a spirometric examination in healthy or affected volunteer subjects in spontaneous breathing or during mechanical ventilation in intubated subjects. It is unknown whether there is a correlation between the velocimetric parameters generated by the Doppler wave with the main ventilatory parameters (Current Volume, Compliance, Plateau pressure, PEEP, Driving pressure constant Tau). There is currently no correlation between B-mode ultrasound pathological patterns with velocimetry data.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Acquisition of Informed Consent

Exclusion Criteria:

* Patients admitted to undergo major thoracic surgery.
* Remote pathological history positive for recurrent PNX (≥ 2), pleural thalking or pleurodesis
* Patients presenting with absolute and relative contraindications to spirometry for1 and 2a patients ie:

recent myocardial infarction (within the past 3 months) or unstable angina hemoptysis thoracic aortic aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients belonging to the operating units involved in the study will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
analyze, by ultrasound examination, the Doppler wave generated by lung sliding and measure the parenchyma sliding velocity | through study completion, an average of 1 year
  The primary purpose of this study is to analyze, by ultrasound examination, the Doppler wave generated by lung sliding and measure the parenchyma sliding velocity in healthy subjects and in patients with established lung disease

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Tonetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna - Anestesiologia e Terapia Intensiva Polivalente
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di Sant'Orsola, UOC Anestesiologia e Terapia Intensiva Polivalente, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, UO Pneumologia, Bologna